CLINICAL TRIAL: NCT02330523
Title: A Prospective, Randomized, Controlled, Multi-center Study With Direct Measure and Histological Evaluation Comparing Xenograft and Allograft for Posterior Buccal Dehiscence Extraction Site Ridge Preservation
Brief Title: An RCT Comparing Xenograft and Allograft for Ridge Preservation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: McGuire Institute (Industry)
Collaborators: Geistlich Pharma AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 13530232
Record Dates: First submitted 2014-12-31; First posted 2015-01-05 (Estimated); Results first posted 2016-02-18 (Estimated); Last update posted 2016-02-18 (Estimated); Status verified 2015-12

CONDITIONS: Tooth Loss
MeSH Terms: conditions — Tooth Loss | interventions — Transplantation, Homologous; Transplantation, Heterologous

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- allograft + x-link collagen membrane (Active Comparator): Demineralized freeze-dried allograft + x-linked collagen membrane will be used for guided bone regeneration of dehiscence buccal defects post extraction.
  Interventions: Device: allograft + x-link collagen membrane
- xenograft + non-x-link collagen (Active Comparator): Xenograft + non-x-linked collagen membrane will be used for guided bone regeneration of dehiscence buccal defects post extraction.
  Interventions: Device: xenograft + non-x-link collagen

INTERVENTIONS:
Device: allograft + x-link collagen membrane — Following resolution of any periodontal issues in the region of study and administration of pre-surgical antibiotic, minimally traumatic extraction with periotomes and flap reflection will be performed. Allograft will be placed according to randomization schedule and in quantity to fill the extraction socket and mimic surrounding ridge dimension. X-link collagen membrane will be trimmed to extend at least 2 mm beyond the margins of the defect, and soft tissue flaps will be re-approximated using resorbable Vicryl® 6-0.
  Arms: allograft + x-link collagen membrane
Device: xenograft + non-x-link collagen — Following resolution of any periodontal issues in the region of study and administration of pre-surgical antibiotic, minimally traumatic extraction with periotomes and flap reflection will be performed. Xenograft will be placed according to randomization schedule and in quantity to fill the extraction socket and mimic surrounding ridge dimension. Non-x-link collagen membrane will be trimmed to extend at least 2 mm beyond the margins of the defect, and soft tissue flaps will be re-approximated using resorbable Vicryl® 6-0.
  Arms: xenograft + non-x-link collagen

SUMMARY:
To compare the effectiveness of demineralized freeze-dried bone allograft + cross-linked collagen membrane with xenograft + non-cross-linked collagen membrane for posterior extraction socket ridge preservation.

DETAILED DESCRIPTION:
Buccal bony wall loss is a common sequela following tooth extraction, and guided bone regeneration (GBR) is a common treatment for the regeneration of ridge form and volume preservation allowing dental implant placement. Many bone augmentation biomaterials are employed to accomplish GBR, and both the medical/ dental community and, subsequently, patients benefit from understanding whether a given GBR biomaterial might be more efficacious. To this end, a randomized, case series comparison of allograft + x-linked collagen membrane versus xenograft + non-x-linked collagen membrane would be beneficial to both the dental community and patients.

The study compares the effectiveness of demineralized freeze-dried bone allograft + x-linked collagen membrane with xenograft + non-x-linked collagen membrane for posterior region extraction socket ridge preservation.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects 18 to 70-yrs of age
2. Subject indicated for posterior tooth extraction (from 1st premolar to 1st molar) intended for implant placement, with adjacent teeth intact (for stent indexing)
3. Subjects with extraction site bony buccal dehiscences at least 1/3 the depth of socket and 1/3 the mesial-distal width of tooth socket
4. Subjects will have read, understood and signed an institutional review board (IRB) approved Informed Consent Form (ICF).
5. Subjects must be able and willing to follow study procedures and instructions.

Exclusion Criteria:

1. Subjects with a history of any tobacco use within the last six months.
2. Subjects with healing disorders (i.e., diabetes mellitus, cancer, HIV, bone metabolic diseases) that could compromise wound healing and/ or preclude implant surgery; or who are currently receiving or have received within two months prior to study entry, systemic corticosteroids, immunosuppressive agents, radiation therapy, and/or chemotherapy which could compromise wound healing and preclude periodontal surgery.
3. Subjects taking intramuscular or intravenous bisphosphonates.
4. Subjects who have a known allergy or sensitivity to alginate, latex, collagen or acrylic.
5. Female subjects who are pregnant or lactating, or who intend to become pregnant during the study duration
6. Subjects participating in other clinical studies involving therapeutic intervention (either medical or dental).
7. Subjects, who in the opinion of the investigator, for any reason other than those listed above, will not be able to complete the study per protocol.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2014-04; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eric T Scheyer, DDS, MS, Principal Investigator — The McGuire Institute
Locations (1):
- Perio Health Professionals, Houston, Texas, United States

REFERENCES:
- [Background] Cook DC, Mealey BL. Histologic comparison of healing following tooth extraction with ridge preservation using two different xenograft protocols. J Periodontol. 2013 May;84(5):585-94. doi: 10.1902/jop.2012.120219. Epub 2012 Jun 9. PMID 22680300

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited at all 9 investigation sites between October 2013 and June 2014.
Groups:
- Allograft + X-link Collagen Membrane: Demineralized freeze-dried allograft + x-linked collagen membrane will be used for guided bone regeneration of dehiscence buccal defects post extraction.
  Guided Bone Regeneration: Following resolution of any periodontal issues in the region of study and administration of pre-surgical antibiotic, minimally traumatic extraction with periotomes and flap reflection will be performed. Test graft materials will be placed according to randomization schedule and in quantity to fill the extraction socket and mimic surrounding ridge dimension. The membranes will be trimmed to extend at least 2 mm beyond the margins of the defect, and soft tissue flaps will be re-approximated using resorbable Vicryl® 6-0.
- Xenograft + Non-x-link Collagen: Xenograft + non-x-linked collagen membrane will be used for guided bone regeneration of dehiscence buccal defects post extraction.
  Guided Bone Regeneration: Following resolution of any periodontal issues in the region of study and administration of pre-surgical antibiotic, minimally traumatic extraction with periotomes and flap reflection will be performed. Test graft materials will be placed according to randomization schedule and in quantity to fill the extraction socket and mimic surrounding ridge dimension. The membranes will be trimmed to extend at least 2 mm beyond the margins of the defect, and soft tissue flaps will be re-approximated using resorbable Vicryl® 6-0.
Period: Overall Study
Arm/Group | Allograft + X-link Collagen Membrane | Xenograft + Non-x-link Collagen
Started | 21 | 19
Completed | 21 | 19
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Allograft + X-link Collagen Membrane | Xenograft + Non-x-link Collagen | Total
Number analyzed (Participants) | 21 | 19 | 40
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.9 (10.7) | 55.3 (13.3) | 55.7 (11.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 9 | 19
  Male | 11 | 10 | 21
Region of Enrollment [Number; unit: participants]
  United States | 21 | 19 | 40

OUTCOME MEASURES:

1. Primary Outcome: Bone Ridge Buccal-Lingual and Apico-Coronal Measures at 6 Months
Description: The primary efficacy parameter will be ridge volume preservation as measured apico-coronal and buccal-lingual using a preformed and marked stent.
Time Frame: Six Months
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Allograft + X-link Collagen Membrane | Xenograft + Non-x-link Collagen
Number analyzed (Participants) | 21 | 19
mm
  Bone Ridge Buccal-Lingual Width | 4.95 (2.65) | 6.71 (2.07)
  Bone Ridge Apico-Coronal Height | 5.29 (3.73) | 6.24 (2.98)

2. Secondary Outcome: New Bone Plus Graft Content at 6-months
Description: New bone and graft content are measured as histomorphometric % vital bone and % mineral (graft remnants) from mid-section bone core biopsies. Histomorphometric analyses are performed with imaging software on composite overview scans. The area of new healing (versus old/ original bony tissues) is demarcated in each section. Within this area, the percentage contributions of each tissue type within the overall area of newly healed tissue is computed, i.e., new bone plus graft content added with connective tissue/ marrow elements totals 100% of the "new healing" area.
Time Frame: Six Months
Measure: Mean (Standard Deviation); unit: percentage of total area
Arm/Group | Allograft + X-link Collagen Membrane | Xenograft + Non-x-link Collagen
Number analyzed (Participants) | 21 | 19
percentage of total area | 46.14 (7.66) | 49.21 (8.27)

3. Secondary Outcome: Wound Closure at 4-weeks
Description: Suture line gap will be measured (buccal-lingual) with a UNC-15 Probe, rounding down to the nearest 0.5 mm.
Time Frame: 4-weeks
Measure: Median (Standard Deviation); unit: mm
Arm/Group | Allograft + X-link Collagen Membrane | Xenograft + Non-x-link Collagen
Number analyzed (Participants) | 21 | 19
mm | 2.26 (2.68) | 0.79 (1.55)

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Allograft + X-link Collagen Membrane | Xenograft + Non-x-link Collagen
Serious Adverse Events (participants affected / at risk) | 0/21 | 0/19
Other Adverse Events (participants affected / at risk) | 1/21 | 0/19
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Allograft + X-link Collagen Membrane (N=21) | Xenograft + Non-x-link Collagen (N=19)
Infection (Infections and infestations) | 1 (1) | 0 (0) — Healing was "as expected" for both treatment modalities; no AEs occurred that could be attributed to the study, though 1 subject presented with a localized infection with suppuration at the test site (DFDBA+RECXC) and was treated with antibiotics.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No